CLINICAL TRIAL: NCT00112931
Title: An Intergroup Randomised Trial of Rituximab Versus a Watch and Wait Strategy in Patients With Advanced Stage, Asymptomatic, Non-Bulky Follicular Lymphoma
Brief Title: Rituximab in Treating Patients With Newly Diagnosed Stage II, Stage III, or Stage IV Follicular Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Cancer Research UK (Other); Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000427312; CRUK-2004-001621-16; EU-20509; ROCHE-CRUK-001621-16
Record Dates: First submitted 2005-06-02; First posted 2005-06-03 (Estimated); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Lymphoma
Keywords: stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Watch and Wait (Active Comparator): Watch and Wait - no treatment
  Interventions: Other: No treatment
- Arm C Rituximab 4 and Rixuximab Maintenance (Experimental): 4 infusions - 375mg/m2 every 2 months. A single dose of rituximab (375mg/m2 will then be given at 12, 20, 28, 36, 44, 52, 60, 68, 76, 84, 92 and 100 weeks
  Interventions: Biological: rituximab

INTERVENTIONS:
Biological: rituximab
  Arms: Arm C Rituximab 4 and Rixuximab Maintenance
Other: No treatment
  Arms: Watch and Wait

SUMMARY:
RATIONALE: Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. It is not yet known whether rituximab is more effective than observation in treating non-Hodgkin's lymphoma.

PURPOSE: This randomized phase III trial is studying rituximab to see how well it works compared to observation in treating patients with newly diagnosed stage II, stage III, or stage IV follicular non-Hodgkin's lymphoma with no symptoms.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare time to initiation of systemic chemotherapy or radiotherapy in patients with newly diagnosed, previously untreated, asymptomatic stage II-IV non-bulky follicular non-Hodgkin's lymphoma treated with rituximab vs observation only.

Secondary

* Compare the frequency of clinical spontaneous remission in patients treated with these regimens.
* Compare overall and cause-specific survival of patients treated with these regimens.
* Determine the effect of rituximab on complete and partial response in patients treated with subsequent systemic chemotherapy.
* Compare quality of life, in terms of functional well-being and anxiety and depression, of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center, disease grade (1 vs 2 vs 3a), disease stage (II vs III vs IV), and age. Patients are randomized to 1 of 3 treatment arms.

* Arm I: Patients undergo observation only until disease progression.
* Arm II: Patients receive induction rituximab IV on day 1. Treatment repeats weekly for up to 4 weeks.
* Arm III: Patients receive induction rituximab as in arm II. Patients then receive maintenance rituximab IV once on day 1 of weeks 12, 20, 28, 36, 44, 52, 60, 68, 76, 84, 92, and 100.

In all arms, treatment continues in the absence of unacceptable toxicity or disease progression requiring systemic chemotherapy* or radiotherapy.

NOTE: *Rituximab administration in arm I is considered initiation of systemic chemotherapy

Quality of life is assessed at baseline (before and after randomization), every 2 months for 2 years, and then every 6 months for 2 years.

Patients are followed every 2 months for 2 years and then every 3 months thereafter.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 600 patients (200 per treatment arm) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed follicular non-Hodgkin's lymphoma

  * Diagnosed within the past 3 months
  * Grade 1, 2, or 3a disease
  * Stage II-IV disease
  * No evidence of histological transformation
* Bidimensionally measurable disease by clinical examination or radiography
* Asymptomatic disease without B symptoms or severe pruritus
* Low tumor burden, defined by all of the following criteria:

  * Lactic dehydrogenase normal
  * Largest nodal or extranodal mass < 7 cm
  * No more than 3 nodal sites with a diameter > 3 cm
  * No clinically detectable significant serous effusion by chest x-ray

    * Clinically non-evident small effusion on CT scan is not considered significant
  * Spleen enlargement ≤ 16 cm by CT scan
* Circulating tumor cells < 5,000/mm^3
* No organ compression (i.e., ureteric obstruction)

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count > 1,500/mm^3
* Platelet count > 100,000/mm^3
* Hemoglobin > 10 g/dL

Hepatic

* AST and ALT normal
* Alkaline phosphatase normal
* Bilirubin normal

Renal

* Creatinine < 2 times upper limit of normal (unless due to lymphoma)

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 12 months after completion of rituximab
* No known HIV positivity
* No other malignancy within the past 2 years except curatively treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No critical organ failure
* No other immediate life-threatening disease

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* No prior therapy for lymphoma

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 462 (Actual)
Dates: Start 2004-09; Primary Completion 2014-03 (Actual); Study Completion 2023-09-14 (Actual)

PRIMARY OUTCOMES:
Time until initiation of therapy (chemotherapy or radiotherapy) | Time from randomisation until the first day systemic chemotherapy or radiotherapy is given. If rituximab is given to patients in the watch and wait arm this will be considered as initiation of chemotherapy.

SECONDARY OUTCOMES:
Frequency of clinical spontaneous remission | From randomisation until the initiation of chemotherapy in the watch and wait arm
Cause specific survival | Time from randomisation to death from lymphoma or immediate therapy related toxicity
Overall survival | Time from randomisation to death from any cause.
Response rate at 25 months | Response at 25 months

CONTACTS AND LOCATIONS:
Overall Officials: Kirit Ardeshna, Study Chair — Mount Vernon Cancer Centre at Mount Vernon Hospital
Locations (72):
- Australia (26):
  - Queen Elizabeth Hospital, Adelaide
  - Royal Adelaide Hospital, Adelaide
  - Ashford Cancer Centre, Black Forest
  - Boxhill Hospital, Box Hill
  - Royal Brisbane and Women's Hospital, Brisbane
  - Canberra Hospital, Canberra
  - Concord Repatriation General Hospital, Concord
  - Frankston Hospital, Frankston
  - Fremantle Hospital, Fremantle
  - Gosford Hospital, Gosford
  - Royal Hobart Hospital, Hobart
  - Nepean Hospital, Kingswood
  - Lismore Base Hospital, Lismore
  - Liverpool Hospital, Liverpool
  - Alfred Hospital, Melbourne
  - Austin Health, Melbourne
  - Peter MacCallum Cancer Centre, Melbourne
  - St Vincent's Hospital, Melbourne
  - Mater Misericordiae Hospital, Newcastle
  - Royal Perth Hospital, Perth
  - Royal North Shore Hospital, St Leonards
  - St Vincent's Hospital, Sydney
  - Westmead Hospital, Westmead
  - Murray Valley Private Hospital, Wodonga
  - Wollongong Hospital, Wollongong
  - Princess Alexandra Hospital, Woolloongabba
- New Zealand (4):
  - Auckland Hospital, Auckland
  - Middlemore Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - North Shore Hospital, Westlake
- United Kingdom (42):
  - Birmingham Heartlands Hospital, Birmingham, England
  - Blackpool Victoria Hospital, Blackpool, England
  - West Suffolk Hospital, Bury St Edmunds, England
  - Kent and Canterbury Hospital, Canterbury, England
  - St. Helier Hospital, Carshalton, England
  - Royal Devon and Exeter Hospital, Exeter, England
  - Queen Elizabeth Hospital, Gateshead, England
  - Medway Maritime Hospital, Gillingham, England
  - Hemel Hempstead General, Hemel Hempstead, England
  - Hull Royal Infirmary, Hull, England
  - West Middlesex University Hospital, Isleworth, England
  - Kettering General Hosptial, Kettering, England
  - Kidderminster Hospital, Kidderminster, England
  - Queen Elizabeth Hospital, Kings Lynn, England
  - Leicester Royal Infirmary, Leicester, England
  - St. George's Hospital, London, England
  - Maidstone Hospital, Maidstone, England
  - Sir James Spence Institute of Child Health at Royal Victoria Infirmary, Newcastle upon Tyne, England
  - Mount Vernon Cancer Centre at Mount Vernon Hospital, Northwood, England
  - Rosemere Cancer Centre at Royal Preston Hospital, Preston, England
  - Alexandra Healthcare NHS, Redditch, England
  - Oldchurch Hospital, Romford, England
  - Pembury Hospital, Royal Tunbridge Wells, England
  - Southampton General Hospital, Southampton, England
  - Staffordshire General Hospital, Stafford, England
  - Royal Marsden - Surrey, Sutton, England
  - Torbay Hospital, Torquay, England
  - Royal Cornwall Hospital, Truro, England
  - Weston General Hospital, Weston-super-Mare, England
  - Worcester Royal Hospital, Worcester, England
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Monklands General Hospital, Airdrie, Scotland
  - Hairmyres Hospital, East Kilbride, Scotland
  - Edinburgh Cancer Centre at Western General Hospital, Edinburgh, Scotland
  - Southern General Hospital, Glasgow, Scotland
  - Raigmore Hospital, Inverness, Scotland
  - Royal Alexandra Hospital, Paisley, Scotland
  - Wishaw General Hospital, Wishaw, Scotland
  - Velindre Cancer Center at Velindre Hospital, Cardiff, Wales
  - Prince Charles Hospital, Merthyr Tydfil, Wales
  - Glan Clwyd Hospital, Rhyl, Wales
  - South West Wales Cancer Institute, Swansea, Wales

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Northend M, Wilson W, Ediriwickrema K, Clifton-Hadley L, Qian W, Rana Z, Martin TL, Townsend W, Young M, Miall F, Cunningham D, Walewski J, Ferhanoglu B, Linton K, Johnston A, Seymour JF, Linch DC, Ardeshna KM. Early rituximab monotherapy versus watchful waiting for advanced stage, asymptomatic, low tumour burden follicular lymphoma: long-term results of a randomised, phase 3 trial. Lancet Haematol. 2025 May;12(5):e335-e345. doi: 10.1016/S2352-3026(25)00034-1. PMID 40306831
- [Derived] Ardeshna KM, Qian W, Smith P, Braganca N, Lowry L, Patrick P, Warden J, Stevens L, Pocock CF, Miall F, Cunningham D, Davies J, Jack A, Stephens R, Walewski J, Ferhanoglu B, Bradstock K, Linch DC. Rituximab versus a watch-and-wait approach in patients with advanced-stage, asymptomatic, non-bulky follicular lymphoma: an open-label randomised phase 3 trial. Lancet Oncol. 2014 Apr;15(4):424-35. doi: 10.1016/S1470-2045(14)70027-0. Epub 2014 Mar 4. PMID 24602760